CLINICAL TRIAL: NCT02409888
Title: Evaluating Interventions for Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Syracuse University (Other); Pacific Institute for Research and Evaluation (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Patrick R. Clifford (PI), Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Pro2013003944; 1R01AA022330-01A1 (NIH)
Record Dates: First submitted 2015-04-01; First posted 2015-04-07 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Motivational Interviewing; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Study participants receive either motivational enhancement therapy (MET) or cognitive behavioral therapy (CBT).
  Interventions: Behavioral: Motivational Enhancement Therapy; Behavioral: Cognitive Behavioral Therapy
- Assessment (Experimental): IB Assessment study participants receive semi-annual assessments specific to their alcohol and other drug use and FC Assessment study participants receive quarterly assessments specific to diverse areas of functioning (e.g., alcohol and other drug use, social, occupational, legal, psychological/psychiatric, marital).
  Interventions: Other: FC Assessment; Other: IB Assessment

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy — The motivational enhancement therapy will be delivered according to the Project MATCH manual.
  Arms: Intervention
Behavioral: Cognitive Behavioral Therapy — The cognitive behavioral therapy will be delivered according to the Project MATCH manual.
  Arms: Intervention
Other: FC Assessment — FC Assessment study participants are exposed to quarterly assessments across broad domains of functioning.
  Arms: Assessment
Other: IB Assessment — IB Assessment study participants are exposed to semi-annual alcohol specific assessments
  Arms: Assessment

SUMMARY:
The purpose of this study is to investigate how behavioral treatments for alcohol use disorders affect behavior change.

ELIGIBILITY:
Inclusion Criteria: Study inclusion criteria are such that study participants must:

1. meet a Diagnostic and Statistical Manual-IV (DSM-IV) alcohol abuse or dependence diagnosis based on the Diagnostic Interview Schedule - IV (DIS-IV);
2. consume a weekly average of at least 24 standard drinks during the baseline period to include at least 5 episodes of heavy drinking;
3. agree not to seek additional alcohol or other substance abuse treatment during the study period;
4. be at least 18 years of age; and
5. be sufficiently proficient in their English speaking ability to interact effectively with the research interviewer.

Exclusion Criteria:

* Individuals assessed as having a drug diagnosis that is more severe than their alcohol diagnosis (e.g., cocaine dependence and alcohol abuse, IV drug use),
* a serious psychiatric diagnosis (e.g., uncontrolled schizophrenia or major depression) as well as those meeting criteria for organic brain impairment, as measured by the mini-mental status examination section of the DIS-IV will be precluded from study participation.

In addition,

* individuals reporting current enrollment in a substance abuse treatment program,
* mandated to substance abuse treatment by a court order, or
* severely socially unstable (e.g., homeless) also will be precluded from study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Alcohol Use | One year post-treatment
  Alcohol use will be measured as percent days abstinent, mean drinks per drinking day, and percent heavy drinking days for study months 3 - 15 (one year post-treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick R Clifford, PhD, Principal Investigator — Rutgers University School of Public Health
Locations (1):
- Rutgers University School of Public Health, New Brunswick, New Jersey, United States